CLINICAL TRIAL: NCT02316756
Title: A Phase 1, Randomized, Double-blind, Sponsor-open, Placebo-controlled First-in-human Trial To Evaluate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Pf-06648671 After Administration Of Single Ascending Doses To Fasted And Fed Healthy Subjects
Brief Title: A Single Ascending Dose Study To Evaluate Safety And Pharmacokinetics Of Compound PF-06648671 In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B7991001; 2014-004394-17 (EudraCT Number)
Record Dates: First submitted 2014-12-10; First posted 2014-12-15 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Healthy Subjects
Keywords: Phase 1, Single-Dose Escalation, Double Blind, Placebo-Controlled, Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, PF-06648671, Plasma Abeta

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Single Ascending Doses Cohort 1 (Experimental): subjects receive 3 active doses and one placebo
  Interventions: Drug: PF-06648671; Drug: Placebo
- Single Ascending Doses Cohort 2 (Experimental): subjects receive 3 doses and one placebo
  Interventions: Drug: PF-06648671; Drug: Placebo
- Cohort 3 (Experimental): optional cohort
  Interventions: Drug: PF-06648671; Drug: Placebo

INTERVENTIONS:
Drug: PF-06648671 — Experimental Pfizer compound which will be dosed as oral suspension
Drug: Placebo — Placebo which will be given as oral suspension

SUMMARY:
This is first in human (FIH), double-blind, sponsor open, placebo-control trial to examine the safety, tolerability, pharmacokinetics and pharmacodynamics following a single ascending doses of PF-06648671 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non childbearing potential
* BMI of 17.5 to 30.5 kg/m2 and a total body weight >50 kg (110 lbs)
* Evidence of a personally signed and dated informed consent document indicating that subject has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drg allergies, but excluding untreated asymptomatic, seasonal allergies at the time of dosing);
* Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study medication (whichever is longer)
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgement of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with AEs and SAEs | 0-6 weeks
  Counts of participants who have TEAEs, defined as newly occuring or worsening after first dose. Relatedness to PF-06648671 will be assessed by the investigator (Yes/No). Participants with multiple occurences of an AE within a category will be counted once within the category
Supine vital sign measurement | 0-6 weeks
  Measurement of blood pressure and pulse rate
Electrocardiogram (ECG) | 0-6 weeks
  Measurement of standard 12-lead ECG, single or triplicate
Number of participants with lab test values of potential clinical importance | 0-6 weeks
  Pre-defined criteria were established for each lab test to identify potential clinical importance

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 0-72 hours post dose
Area Under the Curve From Time Zeor to Last Quantifiable Concentration (AUClast) | 0-72 hours post dose
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) | 0-72 hours post dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0-72 hours post dose
Plasma Decay Half-life (t1/2) | 0-72 hours post dose
Apparent Oral Clearance (CL/F) | 0-72 hours post dose
Apparent Volume of Distribution (Vz/F) | 0-72 hours post dose
Plasma Cmax ratio under fed vs fasted conditions | 0-72 hours post dose
Plasma AUClast ratio under fed vs fasted condition | 0-72 hours post dose
Plasma AUCinf ratio under fed vs fasted conditions | 0-72 hours post dose
Plasma Abeta42 Maximum change from baseline | 0-72 hours post dose
Plasma Abeta42, Area Under the Effect Curve from Time Zero to Last Quantifiable Concentration (AUEC) | 0-72 hours post dose
Plasma Abeta42, Time to Reach Maximum Observed Effect (Tmax) | 0-72 hours post-dose
Plasma Abeta40 Maximum change from baseline | 0-72 hours post dose
Plasma Abeta40, Area Under the Effect Curve from Time Zero to Last Quantifiable Concentration (AUEC) | 0-72 hours post dose
Plasma Abeta40, Time to Reach Maximum Observed Effect (Tmax) | 0-72 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer; Laure Mendes da Costa, MD, Principal Investigator — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

REFERENCES:
- [Derived] Ahn JE, Carrieri C, Dela Cruz F, Fullerton T, Hajos-Korcsok E, He P, Kantaridis C, Leurent C, Liu R, Mancuso J, Mendes da Costa L, Qiu R. Pharmacokinetic and Pharmacodynamic Effects of a gamma-Secretase Modulator, PF-06648671, on CSF Amyloid-beta Peptides in Randomized Phase I Studies. Clin Pharmacol Ther. 2020 Jan;107(1):211-220. doi: 10.1002/cpt.1570. Epub 2019 Sep 11. PMID 31314925